CLINICAL TRIAL: NCT02939404
Title: Energy Intake Response to Short-Term Alterations of Energy Expenditure in Humans
Brief Title: Food Intake Response to Short-Term Modifications of Metabolism in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 999917004; 17-DK-N004 (Other: NIDDK)
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2024-07-03

CONDITIONS: Healthy Volunteers
Keywords: Energy Intake; Energy Expenditure; Eating Behavior; Cold Exposure; Natural History
MeSH Terms: conditions — Feeding Behavior | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 1. Chamber at 24C, fixed diet (Experimental): Chamber at room temperature (24C) with a fixed eucaloric diet
  Interventions: Other: Normal temperature; Other: Fixed diet
- 2. Chamber at 24C, ad libitum diet (Experimental): Chamber at room temperature (24C) with an ad libitum diet (self-select how much food they wish to eat)
  Interventions: Other: Normal temperature; Other: Ad libitum diet
- 3. Chamber at 19C, fixed diet (Experimental): Chamber at cold temperature (16C) with a fixed eucaloric diet
  Interventions: Other: Cold exposure; Other: Fixed diet
- 4. Chamber at 19C, ad libitum diet (Experimental): Chamber at cold temperature (19C) with an ad libitum diet (self-select how much food they wish to eat)
  Interventions: Other: Cold exposure; Other: Ad libitum diet
- 5. Chamber at 24C, fasting (Experimental): Chamber at room temperature (24C) fasting while in chamber and 12 hours before
  Interventions: Other: Normal temperature; Other: Fasting

INTERVENTIONS:
Other: Cold exposure — 23.25 hours inside respiratory chamber with the temperature set to19°C
  Arms: 3. Chamber at 19C, fixed diet; 4. Chamber at 19C, ad libitum diet
Other: Normal temperature — 23.25 hours inside respiratory chamber with the temperature set to 24°C
  Arms: 1. Chamber at 24C, fixed diet; 2. Chamber at 24C, ad libitum diet; 5. Chamber at 24C, fasting
Other: Fixed diet — A diet that matches the participant's caloric needs
  Other Names: Eucaloric diet
  Arms: 1. Chamber at 24C, fixed diet; 3. Chamber at 19C, fixed diet
Other: Ad libitum diet — Participants can eat as much as they want
  Arms: 2. Chamber at 24C, ad libitum diet; 4. Chamber at 19C, ad libitum diet
Other: Fasting — Participants do not eat for 12 hours before and 24 hours in chamber
  Arms: 5. Chamber at 24C, fasting

SUMMARY:
One reason people gain weight is eating more calories from food than what they need for energy over 24 hours. Metabolism is the amount of energy a person uses over 24 hours. Researchers want to study the relationship between changes in metabolism and how much a person eats.

Objectives:

To see how much food a person eats when the body's temperature is cooled. To study how changes in metabolism may alter the amount of food a person eats.

Eligibility:

Healthy people ages 18-55.

Design:

Participants will stay at NIH for 20 days.

During the first 4 days, participants will have:

* Medical exam
* Electrocardiogram
* Blood and urine tests. One blood test includes drinking a sugar solution.
* DXA body composition scan
* Questions about foods they like, physical activity, and personal behavior
* Exercise test on a stationary bicycle

Participants will spend 24-hour periods in a metabolic chamber. The chamber will be at normal room temperature or cooler.

Some times, participants will eat a diet that matches their daily needs (fixed or eucaloric). Other times, they can eat as much as they wish from a vending machine (ad libitum).

Participants will have blood and urine collected.

Participants will swallow an ingestible wireless sensor and wear a small data recorder device.

On the second to last day, participants will stay in the metabolic chamber but only consume water and non-caffeinated sugar-free beverages.

Participants will come back for 1-day visits at six months and one year from the first admission. They will have blood and urine tests, and a DXA scan. They will answer questions on physical activity and food habits.

DETAILED DESCRIPTION:
More than 30% of adults are considered overweight. In general, lifestyle changes (diet and exercise) or current weight loss drugs only lead to about 5 to 10% weight loss. This may be because a person's energy expenditure, aka the number of calories the body uses, leads to hunger and may increase the amount of food a person eats. Cold exposure is known to increase metabolism but it may not lead to weight loss if appetite and the desire for food are also increased. The primary goal of this study is to evaluate whether changing energy expenditure by cool temperature exposure results in changes in food intake. This study will involve a stay on our clinical research unit where we will determine the energy requirements (at 24 degree C) of 68 healthy, adult volunteers without evidence of diabetes. Exposure to cool temperatures (19 degree C) will be used to increase the number of calories a person's body uses in a day. Participants will spend 24 hours in a room that measures energy expenditure while the temperature in the room is turned down, once with a fixed diet (eucaloric) and once with a buffet of food choices (ad libitum). After the fixed diet, volunteers will self-select how much food they wish to eat for one day from a vending machine. Volunteers will also spend one day fasting followed by a day self-selecting their food from the vending machine. Findings from this study will provide knowledge about a possible causal link between energy expenditure and eating behavior. This information may shed light on why many weight loss interventions that increase energy expenditure do not work as well as expected, and may eventually lead to new weight loss approaches and therapies.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Premenopausal women and men <55 years of age
* Body weight <204 kg (<450 pounds) and >= 36 kg (>= 80 pounds)
* Stable weight (+/-5% within past 6 months) as determined by volunteer report
* Healthy, as determined by medical history, physical examination, and laboratory tests

EXCLUSION CRITERIA:

* Age <18 years
* Weight greater than or equal to 204 kg (greater than or equal to 450 pounds, maximum weight of the iDXA machine as per manufacturer s manual), or weight <36 kg (<80 pounds, minimum weight allowed based on the NIH guidelines of blood drawing for research purposes)
* Use of medications affecting metabolism and appetite in the last three months
* Expresses unwillingness to consume all food given during the weight maintaining diet portions of the study (e.g., due to strict dietary restrictions including allergies or vegetarian or kosher diet)
* Current use of tobacco products, marijuana, amphetamines, cocaine, or intravenous drug use
* Current pregnancy, pregnancy within the past 6 months or lactation
* History or clinical manifestation of:

  * Type 1 and Type 2 diabetes mellitus
  * History of surgery for the treatment of obesity
  * Endocrine disorders, such as Cushing s disease, pituitary disorders, and hypo and hyperthyroidism
  * Pulmonary disorders, including chronic obstructive pulmonary disease
  * Cardiovascular diseases, including coronary heart disease, heart failure, arrhythmias, and peripheral artery disease
  * High blood pressure by sitting blood pressure measurement using an appropriate cuff higher than 140/90 mmHg on two or more occasions, or current antihypertensive therapy
  * Liver disease, including cirrhosis, active hepatitis B or C, and AST or ALT greater than or equal to 2x normal
  * Gastrointestinal disease including Crohn s disease, ulcerative colitis, celiac disease or other malabsorptive disorders
  * Abnormal kidney function (eGFR <60 mL/min/1.73m(2))
  * Central nervous system disease, including previous history of cerebrovascular accidents, dementia, neurodegenerative disorders or history of severe head trauma
  * Cancer requiring treatment in the past five years, except for nonmelanoma skin cancers or cancers that have clearly been cured
  * Infectious disease such as active tuberculosis, HIV (by self report), chronic coccidiomycoses or other chronic infections that might influence EE and weight
  * Diagnosis of binge eating disorder, anorexia and major psychiatric disorders based upon the DSM-IV including depression, schizophrenia and psychosis, which may impact the ability of the participant to be in the respiratory chamber for 24 hour time periods
* Chronic ethanol use (more than 3 drinks/day)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Chang, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Unlu Y, Piaggi P, Stinson EJ, De Baca TC, Rodzevik TL, Walter M, Fry H, Krakoff J, Chang DC. Cold induces increased ad libitum energy intake independent of changes in energy expenditure: a controlled crossover trial in adults. Am J Clin Nutr. 2025 Feb;121(2):293-303. doi: 10.1016/j.ajcnut.2024.12.013. Epub 2024 Dec 14. PMID 39675563
- [Derived] Hollstein T, Heinitz S, Ando T, Rodzevik TL, Basolo A, Walter M, Chang DC, Krakoff J, Piaggi P. Metabolic Responses to 24-Hour Fasting and Mild Cold Exposure in Overweight Individuals Are Correlated and Accompanied by Changes in FGF21 Concentration. Diabetes. 2020 Jul;69(7):1382-1388. doi: 10.2337/db20-0153. Epub 2020 Apr 27. PMID 32341039
- [Derived] Hollstein T, Basolo A, Ando T, Votruba SB, Walter M, Krakoff J, Piaggi P. Recharacterizing the Metabolic State of Energy Balance in Thrifty and Spendthrift Phenotypes. J Clin Endocrinol Metab. 2020 May 1;105(5):1375-92. doi: 10.1210/clinem/dgaa098. PMID 32118268

RESULTS

PARTICIPANT FLOW:
Groups:
- Chamber at 19°C With Fixed Diet First: Order of chambers will be Chamber at normal room temperature (24°C) with fixed eucaloric diet, Chamber at 24°C with ad libitum diet, Chamber at 19°C with fixed eucaloric diet, Chamber at 19°C with ad libitum diet, and Chamber at 24°C fasting.
  Normal room temperature: 23.25 hours inside respiratory chamber with the temperature set to 24°C
  Fixed diet: A diet that matches the participant's caloric needs
  Ad libitum diet: Participants can eat as much as they want (self-select how much food they wish to eat)
- 2. Chamber at 19°C, ad Libitum Diet First: Order of chambers will be Chamber at normal room temperature (24°C) with fixed eucaloric diet, Chamber at 24°C with ad libitum diet, Chamber at 19°C with ad libitum diet, Chamber at 19°C with fixed eucaloric diet, and Chamber at 24°C fasting.
  Normal room temperature: 23.25 hours inside respiratory chamber with the temperature set to 24°C
  Fixed diet: A diet that matches the participant's caloric needs
  Ad libitum diet: Participants can eat as much as they want (self-select how much food they wish to eat)
Period: Chamber at 24°C, Fixed Diet
Arm/Group | Chamber at 19°C With Fixed Diet First | 2. Chamber at 19°C, ad Libitum Diet First
Started | 24 | 30
Completed | 19 | 27
Not Completed | 5 | 3
Period: Chamber at 24°C, ad Libitum Diet
Arm/Group | Chamber at 19°C With Fixed Diet First | 2. Chamber at 19°C, ad Libitum Diet First
Started | 24 | 30
Completed | 19 | 27
Not Completed | 5 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 3 | 2
Period: Chamber at 19°C, Fixed Diet
Arm/Group | Chamber at 19°C With Fixed Diet First | 2. Chamber at 19°C, ad Libitum Diet First
Started | 24 | 30
Completed | 19 | 27
Not Completed | 5 | 3
Period: Chamber at 19°C, ad Libitum Diet
Arm/Group | Chamber at 19°C With Fixed Diet First | 2. Chamber at 19°C, ad Libitum Diet First
Started | 24 | 30
Completed | 19 | 27
Not Completed | 5 | 3
Period: Chamber at 24°C, Fasting
Arm/Group | Chamber at 19°C With Fixed Diet First | 2. Chamber at 19°C, ad Libitum Diet First
Started | 24 | 30
Completed | 19 | 27
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chamber at 19°C With Fixed Diet First | 2. Chamber at 19°C, ad Libitum Diet First | Total
Number analyzed (Participants) | 24 | 30 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (9.4) | 37.8 (10.9) | 36.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 14 | 18 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 14 | 19 | 33
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 2 | 2 | 4
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: 24-hour Energy Expenditure (kcal)
Description: Energy expenditure (EE) as measured during 24 hours in a whole-room calorimeter
Time Frame: Days 6 (Chamber at 24°C, fixed diet), 10(Chamber at 24°C, ad libitum diet), 14(Chamber at 19°C, fixed or ad libitum diet), 18(Chamber at 19°C, fixed or ad libitum diet), and 21(Chamber at 24°C, fasting)
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Chamber at 19°C With Fixed Diet First | 2. Chamber at 19°C, ad Libitum Diet First
Number analyzed (Participants) | 18 | 27
kcal
  Chamber at 24°C, fixed diet | 2256 (393) | 2166 (302)
  Chamber at 24°C, ad libitum diet | 2563 (422) | 2487 (385)
  Chamber at 19°C, fixed diet | 2271 (360) | 2153 (304)
  Chamber at 19°C, ad libitum diet | 2552 (418) | 2505 (401)
  Chamber at 24°C, fasting | 2135 (337) | 1998 (296)

2. Primary Outcome: 24-hour Energy Intake (kcal)
Description: Energy intake as measured during 24 hours in a whole-room calorimeter
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Chamber at 19°C With Fixed Diet First | 2. Chamber at 19°C, ad Libitum Diet First
Number analyzed (Participants) | 18 | 27
kcal
  Chamber at 24°C, fixed diet | 3811 (1140) | 3694 (1503)
  Chamber at 24°C, ad libitum diet | 4091 (1054) | 4359 (1404)
  Chamber at 19°C, fixed diet | 4014 (1136) | 4075 (1587)
  Chamber at 19°C, ad libitum diet | 4509 (1255) | 4762 (1610)
  Chamber at 24°C, fasting | 3795 (1223) | 4112 (1406)

3. Secondary Outcome: 24- Hour Respiratory Quotient (RQ)
Description: RQ, an approximation for the ratio of carbohydrate-to-fat oxidation rates, is measured while in the chamber
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Chamber at 19°C With Fixed Diet First | 2. Chamber at 19°C, ad Libitum Diet First
Number analyzed (Participants) | 18 | 27
ratio
  Chamber at 24°C, fixed diet | 0.868 (0.024) | 0.868 (0.029)
  Chamber at 24°C, ad libitum diet | 0.925 (0.056) | 0.935 (0.06)
  Chamber at 19°C, fixed diet | 0.872 (0.02) | 0.867 (0.032)
  Chamber at 19°C, ad libitum diet | 0.909 (0.037) | 0.916 (0.045)
  Chamber at 24°C, fasting | 0.793 (0.022) | 0.789 (0.03)

4. Secondary Outcome: Leptin
Description: Plasma leptin (ng/ml)
Time Frame: Days 6 (Chamber at 24°C, fixed diet), 14(Chamber at 19°C, fixed diet) or 18(Chamber at 19°C, fixed diet), and 21(Chamber at 24°C, fasting)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Chamber at 19°C With Fixed Diet First | 2. Chamber at 19°C, ad Libitum Diet First
Number analyzed (Participants) | 18 | 27
ng/mL
  Chamber at 24°C, fixed diet | 26.1 (26.4) | 26.5 (30.5)
  Chamber at 19°C, fixed diet | 29.5 (30.1) | 27.8 (30.3)
  Chamber at 24°C, fasting | 18.3 (19.9) | 16.6 (22.1)

5. Secondary Outcome: Secretin
Description: Plasma secretin (ng/ml)
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Chamber at 19°C With Fixed Diet First | 2. Chamber at 19°C, ad Libitum Diet First
Number analyzed (Participants) | 18 | 27
ng/mL
  (Chamber at 24°C, fixed diet | 0.91 (0.22) | 0.91 (0.25)
  (Chamber at 19°C, fixed diet | 1.03 (0.26) | 1.00 (0.25)
  (Chamber at 24°C, fasting | 0.99 (0.24) | 1.01 (0.24)

6. Secondary Outcome: Ghrelin
Description: Plasma grehlin (pg/ml)
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Chamber at 19°C With Fixed Diet First | 2. Chamber at 19°C, ad Libitum Diet First
Number analyzed (Participants) | 18 | 27
pg/mL
  Chamber at 24°C, fixed diet | 502 (254) | 644 (274)
  Chamber at 19°C, fixed diet | 544 (277) | 605 (311)
  Chamber at 24°C, fasting | 575 (293) | 581 (304)

7. Secondary Outcome: FGF-21
Description: Plasma FGF-21 (pg/ml)
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Chamber at 19°C With Fixed Diet First | 2. Chamber at 19°C, ad Libitum Diet First
Number analyzed (Participants) | 18 | 27
pg/mL
  Chamber at 24°C, fixed diet | 94 (73) | 98 (72)
  Chamber at 19°C, fixed diet | 98 (81) | 113 (90)
  Chamber at 24°C, fasting | 106 (66) | 108 (76)

8. Secondary Outcome: Core Body Temperature (C)
Description: Core body temperature measured in chamber
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: C
Arm/Group | Chamber at 19°C With Fixed Diet First | 2. Chamber at 19°C, ad Libitum Diet First
Number analyzed (Participants) | 10 | 21
C
  Chamber at 24°C, fixed diet | 36.98 (0.15) | 37.02 (0.17)
  Chamber at 19°C, fixed diet | 36.97 (0.19) | 36.95 (0.20)
  Chamber at 24°C, fasting | 36.98 (0.21) | 36.98 (0.21)

9. Secondary Outcome: Weight Change at 6 Months
Description: Weight change from baseline to 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Chamber at 19°C With Fixed Diet First | 2. Chamber at 19°C, ad Libitum Diet First
Number analyzed (Participants) | 7 | 11
kg | 0.3 (5.6) | -0.5 (8.1)

10. Secondary Outcome: Weight Change at 12 Months
Description: Weight change from baseline to 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Chamber at 19°C With Fixed Diet First | 2. Chamber at 19°C, ad Libitum Diet First
Number analyzed (Participants) | 6 | 11
kg | 1.0 (8.9) | -0.6 (8.9)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Chamber at 19°C With Fixed Diet First | 2. Chamber at 19°C, ad Libitum Diet First
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/30
Other Adverse Events (participants affected / at risk) | 2/24 | 1/30
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chamber at 19°C With Fixed Diet First (N=24) | 2. Chamber at 19°C, ad Libitum Diet First (N=30)
Gastroesophageal reflux disease symptoms at Chamber at 24°C, fixed diet (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastroesophageal reflux disease symptoms at Chamber at 19°C, fixed diet (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT02939404/Prot_SAP_000.pdf